CLINICAL TRIAL: NCT00693030
Title: In-Vivo Vascular Response of Sirolimus-,Paclitaxel- and Zotarolimus-Eluting Stents in Long Lesions Requiring Overlapping. A Prospective, Randomized, Controlled Study Using Optical Coherence Tomography
Brief Title: Optical Coherence Tomography for Drug Eluting Stent Safety
Acronym: ODESSA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Case Western Reserve University (Other); Medtronic Vascular (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Giulio Guagliumi, Cardiovascular Department Ospedali Riuniti di Bergamo ITALY
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0106
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Percutaneous Coronary Interventions; Drug-Eluting stents; Optical Coherence Tomography; Thrombosis; Long lesions in native vessel requiring stents in overlap
MeSH Terms: conditions — Coronary Artery Disease; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Device, Sirolimus drug-eluting stents implanted in overlap
  Interventions: Device: sirolimus drug eluting coronary stent Cypher™ (Cordis Corp, Johnson & Johnson Co)
- 2 (Active Comparator): Device, paclitaxel polymer drug eluting stent
  Interventions: Device: paclitaxel polymer drug eluting stent Taxus Libertè™ (Boston Scientific, Natick MS)
- 3 (Active Comparator): Device, zotarolimus drug eluting stent
  Interventions: Device: zotarolimus drug eluting coronary stent Endeavor™ (Medtronic, Santa Rosa, CA)
- 4 (Active Comparator): bare metal coronary stents
  Interventions: Device: Libertè bare metal coronary stent Libertè™ BMS(Boston Scientific, Natick, MS)

INTERVENTIONS:
Device: sirolimus drug eluting coronary stent Cypher™ (Cordis Corp, Johnson & Johnson Co) — comparison of multiple drug eluting stents
  Other Names: Cypher™ (Cordis Corp, Johnson & Johnson Co) DES
  Arms: 1
Device: paclitaxel polymer drug eluting stent Taxus Libertè™ (Boston Scientific, Natick MS) — comparison of multiple drug eluting coronary stents
  Other Names: Taxus Libertè™ (Boston Scientific, Natick MS) DES
  Arms: 2
Device: zotarolimus drug eluting coronary stent Endeavor™ (Medtronic, Santa Rosa, CA) — comparison of multiple drug eluting coronary stents
  Other Names: Endeavor™ (Medtronic, Santa Rosa, CA) DES
  Arms: 3
Device: Libertè bare metal coronary stent Libertè™ BMS(Boston Scientific, Natick, MS) — comparison of DES in overlap vs BMS in overlap
  Other Names: Libertè™ BMS(Boston Scientific, Natick, MS)
  Arms: 4

SUMMARY:
Increasing lesion complexity in percutaneous coronary interventions (PCI) has warranted the use of overlapping drug-eluting stents. Whether the substantial impairment of arterial healing observed at sites of overlap in preclinical pathologic studies persists in patients undergoing PCI is unknown. Consecutive patients with long lesions in native coronary vessels requiring stents in overlap are prospectively randomized to receive multiple sirolimus-,paclitaxel polymer-or zotarolimus eluting stents versus bare metal stents. The completeness of stent struts coverage and/or late malapposition are evaluated by Optical Coherence Tomography at 6 months follow-up

DETAILED DESCRIPTION:
If overlapping drug-eluting stents provide increased vessel toxicity is not known. Given the association of delayed healing and incomplete endothelialization observed in animal and human autopsy studies at overlapping sites it is unclear why most patients do well with multiple DES implanted. OCT detecs smaller degrees of in-stent neointima more accurately than IVUS and might be a useful method for identify strut coverage and/or malapposition.

Patients if eligible on the basis of clinical and angiographic criteria, are randomized (2:2:2:1) to receive multiple TAXUS Libertè™ vs Cypher Select™ vs Endeavor™ vs Libertè BM stents, in overlap. Stent implantation are done accordingly to the normal interventional practice. QCA and IVUS are performed at the end of optimal stents placement per visual judgement (residual stenosis < 10%, TIMI 3 flow). Stent, lumen size and volume as well as complete stent strut apposal will be determined by IVUS analysis. Clinical follow-up will take place at 1 month (±1 week), 6 months (±2 weeks) and 1 year (±2 weeks). At 6-months follow-up all patients will undergo a quantitative coronary angiography (QCA), IVUS and Optical Coherence Tomography (LightLab OCT Imaging M2, automated pull back and flushing combination)assessments.

OCT images will be acquired at 15-30 frames per second. Blind corelab quantitative strut by strut analysis will be performed using a novel dedicated software at each 0.5 mm section. The following OCT variables will be evaluated:number of visualized strut per section, mean-max neointimal thickness per section, % struts well apposed with neointima at overlapping vs non overlapping sites, % struts without neointima, % struts malapposed, rate of > 30% uncovered struts/total number of struts per section.

ELIGIBILITY:
Inclusion Criteria:

1. Native coronary artery disease with ≥ 75% diameter stenosis
2. Lesion length ≥ 20 mm,
3. Vessel size in between 2.5 and 3.5 mm.
4. Multiple, overlapped DES vs BMS placement (intention to overlap ≥ 4 mm)
5. Signed patient informed consent

Exclusion Criteria:

1. left main coronary artery disease,
2. lesions in coronary artery bypass grafts,
3. acute myocardial infarction,
4. poor cardiac function as defined by left ventricular global ejection fraction ≤ 30%.
5. allergy to aspirin and or clopidogrel/ticlo,
6. renal failure with creatinine value > 2.5,
7. no suitable anatomy for OCT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-06 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Number of uncovered and/or malapposed stent struts at overlapping versus non overlapping sites in drug eluting vs bare metal stents | 6 months

SECONDARY OUTCOMES:
Ischemia Driven Target Vessel Failure | 12 months
Number of uncovered and/or malapposed stent struts at overlapping sites in sirolimus-, paclitaxel- or zotarolimus eluting stents | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Guagliumi, MD, Principal Investigator — Cardiovascular Department Ospedali Riuniti di Bergamo
Locations (1):
- Cardiovascular Department Ospedali Riuniti di Bergamo, Bergamo, Italy

REFERENCES:
- [Background] Joner M, Finn AV, Farb A, Mont EK, Kolodgie FD, Ladich E, Kutys R, Skorija K, Gold HK, Virmani R. Pathology of drug-eluting stents in humans: delayed healing and late thrombotic risk. J Am Coll Cardiol. 2006 Jul 4;48(1):193-202. doi: 10.1016/j.jacc.2006.03.042. Epub 2006 May 5. PMID 16814667
- [Background] Finn AV, Kolodgie FD, Harnek J, Guerrero LJ, Acampado E, Tefera K, Skorija K, Weber DK, Gold HK, Virmani R. Differential response of delayed healing and persistent inflammation at sites of overlapping sirolimus- or paclitaxel-eluting stents. Circulation. 2005 Jul 12;112(2):270-8. doi: 10.1161/CIRCULATIONAHA.104.508937. Epub 2005 Jul 5. PMID 15998681
- [Background] Finn AV, Joner M, Nakazawa G, Kolodgie F, Newell J, John MC, Gold HK, Virmani R. Pathological correlates of late drug-eluting stent thrombosis: strut coverage as a marker of endothelialization. Circulation. 2007 May 8;115(18):2435-41. doi: 10.1161/CIRCULATIONAHA.107.693739. Epub 2007 Apr 16. PMID 17438147
- [Background] Finn AV, Nakazawa G, Joner M, Kolodgie FD, Mont EK, Gold HK, Virmani R. Vascular responses to drug eluting stents: importance of delayed healing. Arterioscler Thromb Vasc Biol. 2007 Jul;27(7):1500-10. doi: 10.1161/ATVBAHA.107.144220. Epub 2007 May 17. PMID 17510464
- [Background] Nakazawa G, Finn AV, John MC, Kolodgie FD, Virmani R. The significance of preclinical evaluation of sirolimus-, paclitaxel-, and zotarolimus-eluting stents. Am J Cardiol. 2007 Oct 22;100(8B):36M-44M. doi: 10.1016/j.amjcard.2007.08.020. PMID 17950831
- [Background] Matsumoto D, Shite J, Shinke T, Otake H, Tanino Y, Ogasawara D, Sawada T, Paredes OL, Hirata K, Yokoyama M. Neointimal coverage of sirolimus-eluting stents at 6-month follow-up: evaluated by optical coherence tomography. Eur Heart J. 2007 Apr;28(8):961-7. doi: 10.1093/eurheartj/ehl413. Epub 2006 Nov 29. PMID 17135281
- [Background] Bouma BE, Tearney GJ, Yabushita H, Shishkov M, Kauffman CR, DeJoseph Gauthier D, MacNeill BD, Houser SL, Aretz HT, Halpern EF, Jang IK. Evaluation of intracoronary stenting by intravascular optical coherence tomography. Heart. 2003 Mar;89(3):317-20. doi: 10.1136/heart.89.3.317. PMID 12591841
- [Background] Takano M, Inami S, Jang IK, Yamamoto M, Murakami D, Seimiya K, Ohba T, Mizuno K. Evaluation by optical coherence tomography of neointimal coverage of sirolimus-eluting stent three months after implantation. Am J Cardiol. 2007 Apr 15;99(8):1033-8. doi: 10.1016/j.amjcard.2006.11.068. Epub 2007 Feb 23. PMID 17437723
- [Background] Yamaguchi T, Terashima M, Akasaka T, Hayashi T, Mizuno K, Muramatsu T, Nakamura M, Nakamura S, Saito S, Takano M, Takayama T, Yoshikawa J, Suzuki T. Safety and feasibility of an intravascular optical coherence tomography image wire system in the clinical setting. Am J Cardiol. 2008 Mar 1;101(5):562-7. doi: 10.1016/j.amjcard.2007.09.116. Epub 2008 Jan 10. PMID 18307999
- [Derived] Guagliumi G, Musumeci G, Sirbu V, Bezerra HG, Suzuki N, Fiocca L, Matiashvili A, Lortkipanidze N, Trivisonno A, Valsecchi O, Biondi-Zoccai G, Costa MA; ODESSA Trial Investigators. Optical coherence tomography assessment of in vivo vascular response after implantation of overlapping bare-metal and drug-eluting stents. JACC Cardiovasc Interv. 2010 May;3(5):531-9. doi: 10.1016/j.jcin.2010.02.008. PMID 20488410